CLINICAL TRIAL: NCT06885619
Title: Prediction of Left Ventricular Adverse Remodeling and Major Adverse Cardiovascular Events in Patients With Acute Myocardial Infarction Though Plasma Multiomics Analysis
Brief Title: Prediction of LVAR and MACE in AMI Though Plasma Multiomics Analysis
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2025013
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-02

CONDITIONS: Acute Myocardial Infarction (AMI); Left Ventricular Remodeling; Major Adverse Cardiovascular Event; Plasma Multi-Omics
MeSH Terms: conditions — Ventricular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples were centrifuged to separate plasma, which was then aliquoted and stored at -80°C for long-term preservation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with AMI: Patients diagnosed with AMI (ST-segment elevation myocardial infarction [STEMI] and non-ST-segment elevation myocardial infarction [NSTEMI])
  Interventions: Other: Diagnostic Test: echocardiography and blood collection

INTERVENTIONS:
Other: Diagnostic Test: echocardiography and blood collection — Blood samples were collected from all patients at the time of myocardial infarction (MI) diagnosis. For those with acute ST-elevation myocardial infarction, blood samples were taken on the day of diagnosis(T0), as well as two days (T1), one week (T2) and one month (T3) after percutaneous coronary intervention (PCI). Echocardiography was performed at the time of STEMI diagnosis, and then again at one week, one month, and six months post-onset.

SUMMARY:
To identify plasma multi-omics biomarkers that predict left ventricular adverse remodeling (LVAR) and major adverse cardiovascular events (MACE) in patients with acute myocardial infarction, and to investigate the molecular pathways linked to LVAR and MACE.

DETAILED DESCRIPTION:
Despite advances in AMI treatment, a substantial proportion of patients develop LVAR, leading to heart failure and increased MACE risk. Conventional biomarkers (e.g., troponin, NT-proBNP) lack sufficient predictive power for adverse outcomes. Multi-omics approaches - integrating proteomics(e.g., exosome proteomics), metabolomics, transcriptomics and lipidomics - offer a systems-level view that may uncover novel prognostic signatures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosis of AMI (STEMI or NSTEMI) confirmed by clinical criteria, electrocardiogram (ECG), and cardiac biomarkers (e.g., troponin).
3. Willingness to provide informed consent.

Exclusion Criteria:

1. Prior surgery or trauma.
2. Renal failure with glomerular filtration <30 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals diagnosed with acute myocardial infarction (MI), selected by the site personnel according to predefined inclusion criteria. The cohort comprises 1,000 patients, whose baseline clinical characteristics and plasma biomarkers will be assessed.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 2025-1-1 to 2027-12-31
  Identify T0 plasma multi-omics biomarkers that predict cardiac death, myocardial infarction, heart failure, and stroke.

SECONDARY OUTCOMES:
adverse cardiac remodeling | 2025-1-1 to 2027-12-31
  To assess the predictive ability of multi-omics biomarkers in T0 plasma for adverse cardiac remodeling, and to identify new candidate markers for forecasting this condition.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Wang, Dr., Principal Investigator — Beijing Anzhen hospital, Capital Mediacl University.; Tanxi Cai, Dr., Study Director — Institute of Biophysics, Chinese Academy of Sciences
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided